CLINICAL TRIAL: NCT03177486
Title: Frank Score and Its Guidance Significance of Making Treatment Strategy in Coronary Artery Disease
Brief Title: Frank Score and Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Shaanxi Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhongwei, Attending doctor, Shaanxi Provincial People's Hospital
Other Study IDs: FrankSyntax
Record Dates: First submitted 2017-05-29; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Disease
Keywords: Syntax score; Frank sign; Coronary angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with coronary artery disease (CAD) were enrolled. CAD was diagnosed by coronary angiography which also resulted Syntax score. Images of left and right ears were captured by a digital camera. Frank score of each patients was calculated based on characteristics and numbers of wrinkles of the earlobes. Statistic analysis were carried out to analyze the correlation between Frank Score and Syntax Score.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis coronary artery disease by coronary angiography

Exclusion Criteria:

* Diagnosis of malignant tumor
* Positive heart transplant history
* Positive CABG history
* Positive PCI history
* Pregnant and lactating women
* Diagnosis of chronic kidney disease
* Any external ear trauma or disease history

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients receiving coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

PRIMARY OUTCOMES:
Syntax score completed | Up to 30 minutes after completion of coronary angiography
  Syntax score is calculated by two experienced cardiologists according to the results of coronary angiography

SECONDARY OUTCOMES:
Follow-up MACE | When MACE is reported or up to 1 year after diagnosis of coronary artery disease
  MACE is reported in follow-up patients

CONTACTS AND LOCATIONS:
Locations (1):
- Shaanxi Provincial People's Hospital, Xi'an, Shaanxi, China